CLINICAL TRIAL: NCT03985969
Title: Phase 1, Open-label Study, in Healthy Male Volunteers to Evaluate the Potential Effect of Indomethacin on the Pharmacokinetics Parameters of Elafibranor
Brief Title: Study to Investigate the Potential Drug-Drug Interaction Between Elafibranor and Indomethacin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: GFT505-119-15; 2019-001451-38 (EudraCT Number)
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Drug-drug Interaction
Keywords: Healthy volunteers; Elafibranor
MeSH Terms: interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid; Indomethacin

STUDY DESIGN:
Intervention Model Description: Open-label, one sequence crossover, single-centre, single group assignment Phase 1 study in healthy male Caucasians volunteers, aged between 18-50 years old (inclusive)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DDI (Experimental): Period 1: study of elafibranor's pharmacokinetics Period 2: study of elafibranor's pharmacokinetics under CHRONO-INDOCID® (indomethacin) at steady state
  Interventions: Drug: elafibranor; Drug: CHRONO-INDOCID

INTERVENTIONS:
Drug: elafibranor — Elafibranor 120mg is a coated tablet for oral administration
  Other Names: GFT505
Drug: CHRONO-INDOCID — CHRONO-INDOCID 75mg is a capsule for bis in die (bid) oral administration
  Other Names: Indomethacin

SUMMARY:
The enzyme responsible for the conversion of elafibranor into its active metabolite, GFT1007, has not been formally identified, but it is believed to have similar characteristics to an α,β-ketoalkene reductase previously identified in rat liver cytosol. In vitro studies in human liver cytosol fractions have shown that indomethacin inhibits the enzyme responsible of the transformation of elafibranor into GFT1007. As a result, indomethacin was included in the list of prohibited co-medications in all clinical trials with elafibranor, and a formal Drug-Drug Interaction (DDI) clinical study is being conducted to elucidate the effect of indomethacin on elafibranor pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for enrolment into the trial:

1. Provide written informed consent prior to the conduct of any study related procedures;
2. Healthy Caucasian male participant, aged between 18 and 50 years (inclusive);
3. Non-smoker participant or smoker of not more than 5 cigarettes a day within one year prior to Inclusion visit;
4. Body Mass Index (BMI) between 19 and 28 kg/m² and Body Weight (BW) not lower than 55 kg at both Screening visit and Inclusion visit;
5. Considered as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination) at both Screening and Inclusion visits. This will include no variation of body weight of more than 5% between screening and inclusion visits;
6. Normal blood pressure (BP) and heart rate (HR) at both Screening and Inclusion visits after 5 minutes in supine position:

90 mmHg ≤ systolic blood pressure (SBP) ≤ 145 mmHg, 50 mmHg ≤ diastolic blood pressure (DBP) ≤ 90 mmHg, 45 bpm ≤ HR ≤ 90 bpm. Out-of-range values that are not clinically significant, as determined by the Investigator, may be repeated twice and the participant may be enrolled if at least 1 repeated value is within the specified ranges; 7. Normal electrocardiogram (ECG) recording on a 12-lead ECG at both Screening and Inclusion visits: 120 ≤ PR < 220 ms, QRS < 110 ms, QTcf ≤ 430 ms. No sign of any trouble of sinusal automatism, or considered as non clinically significant by the Investigator.

Out-of-range values that are not clinically significant (as determined by the Investigator) may be repeated twice during Screening and Inclusion visits, and the participant may be enrolled if at least 1 repeated value is within the specified normal ranges; 8. Laboratory parameters within the normal range of the laboratory (haematological, blood chemistry tests, urinalysis) at Screening and Inclusion visits. Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator; 9. Participant with normal dietary habits; 10. Covered by Health Insurance System and in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

Participants presenting with any of the following criteria will not be included in the trial:

1. Any history or presence of significant cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic or infectious disease or malignant tumor. Specific attention should be paid for history or presence of any hemorrhage/ulceration of the GI tract;
2. Evidence or history of gastrointestinal, hepatic, or renal disease, surgery or resection that would potentially alter absorption, distribution, metabolism, or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed. Bariatric surgery will not be allowed;
3. Major surgery within 28 days prior to screening or major surgery planned within 6 months following participation to the study;
4. Frequent headaches (>2 times /month) and / or migraine, recurrent nausea and / or vomiting;
5. Symptomatic hypotension at both Screening and Inclusion visits, whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP (≥20mmHg) or DBP (≥10mmHg) within three minutes when changing from the supine to the standing position;
6. Blood donation (including in the frame of a clinical trial) within 2 months before administration or blood donation planned during the study or within 2 months following participation to the study;
7. Receipt of blood products within 2 months prior to Inclusion visit;
8. General anesthetics within the 3 months prior to first administration;
9. History or presence of any allergy or unusual reactions to drugs or anesthetics or known hypersensibility to the investigational products (elafibranor and/or CHRONO-INDOCID®) or their excipients;
10. Any medication that may interfere with study medications absorption, distribution, metabolism or excretion or could lead to induction or inhibition of microsomial enzymes within 3 months prior to first administration;
11. Any drug intake (except paracetamol 3g/d) during the last month prior to inclusion;
12. A positive alcohol test result or urine screen for drugs of abuse result at Screening or Inclusion visits;
13. Any history or suspicion of consumption of any drug of abuse (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, methamphetamines, methadone, methylenedioxymethamphetamine (MDMA), opiates, tricyclic antidepressant) or alcohol (alcohol consumption > 40 grams/day), from Screening to end of the study;
14. Consumption of nutritional supplements, herb-containing drug preparations (including Chinese medicines) or other foods or beverages (e.g., grapefruit and xanthine-containing foods or beverages) that may affect drug-metabolizing enzymes or transporters within 48 hours before Inclusion visit and until end of study visit;
15. Positive for hepatitis B or hepatitis C, or positive results for HIV 1 or 2 tests;
16. Participant unable to abstain from intensive muscular effort;
17. Participant who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development;
18. Participant in the exclusion period of a previous study;
19. Participant who, considering the indemnities of the present study, would have received more than 4500 Euros for his participation in biomedical research within the 12 last months, including the indemnities for the present study;
20. Participant who cannot be contacted in case of emergency;
21. Participant with no legal capacity or limited legal capacity or unable to give an informed consent.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males are eligible
Enrollment: 26 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetics: Area under curve from dosing time to infinity (AUC(0-∞)) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of elafibranor
Plasma pharmacokinetics: Maximum plasma drug concentration (Cmax) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of elafibranor

SECONDARY OUTCOMES:
Plasma pharmacokinetics: Area under curve from dosing time to infinity (AUC(0-∞)) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of GFT1007
Plasma pharmacokinetics: Maximum plasma drug concentration (Cmax) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of GFT1007

OTHER OUTCOMES:
Plasma pharmacokinetics: Area under curve from dosing time to last measurement (AUC(0-t)) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of elafibranor and GFT1007
Plasma pharmacokinetics: Elimination half-life (t1/2) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of elafibranor and GFT1007
Plasma pharmacokinetics: Time of maximum observed concentration (tmax) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of elafibranor and GFT1007
Plasma pharmacokinetics: Area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total area under the plasma concentration-time curve (%AUCextra) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of elafibranor and GFT1007
Plasma pharmacokinetics: Apparent total clearance (CL/F) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of elafibranor
Plasma pharmacokinetics: Apparent volume of distribution (Vd/F) | Pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose (336 and 384 hours post-dose added in sequence 2)
  of elafibranor

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Birman, MD, Study Director — Genfit
Locations (1):
- Eurofins Optimed Clinical Pharmacology Unit, Gières, France

IPD SHARING:
Plan to Share IPD: No